CLINICAL TRIAL: NCT06256250
Title: The Effect of Different Instrumentation Techniques on the Post-Operative Pain in Pulpectomy Treatment of Primary Molars: A Blind Randomized Controlled Clinical Trial
Brief Title: Assessment of Post-operative Pain After Different Instrumentation Techniques in Pulpectomy Treatment of Primary Molars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amal Taha, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0106023PP
Record Dates: First submitted 2023-12-11; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pulp Necroses
Keywords: pulpectomy, XP endo shaper, post operative pain
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- group (1): the adaptive xp endo shaper (Experimental): the root canals of primary molars will be cleaned and shaped in pulpectomy treatment using the adaptive xp endo shaper. it is single file technique saves time and help with patient cooperation.
  Interventions: Procedure: pulpectomy treatment will be done using the adaptive xp endo shaper.
- group (2): Fanta AF baby file (Experimental): the root canals of primary molars will be cleaned and shaped in pulpectomy treatment using FANTA AF baby files. it is pediatric rotary system consists of 4 files specialized for primary molars.
  Interventions: Procedure: pulpectomy treatment will be done using FANTA AF baby files.
- group (3): hand k files (Active Comparator): the root canals of primary molars will be cleaned and shaped in pulpectomy treatment using hand k files. they are manual files, they are standard for root canal treatment (control group)
  Interventions: Procedure: pulpectomy treatment will be done using hand k files.

INTERVENTIONS:
Procedure: pulpectomy treatment will be done using the adaptive xp endo shaper. — the patient will be anesthetized by local anesthesia. the rubber dam will be used for isolation. caries will be removed using high speed handpiece. determination of working length using apex locator. the canal patency will be checked with a # 10 K file, and gliding path until #15 K- file. the root canals of primary molars will be cleaned and shaped in pulpectomy treatment using the adaptive xp endo shaper. it is single file technique saves time and help with patient cooperation . the endomotor will be activated at aspeed of 800 rpm and 1 Ncm torque. the canals will be irrigated using 2.5% Nacol ending with 0.9% normal saline canal irrigation. the canals will be dried with paper points and obturated with Metapex. teeth will be restored by glass ionomer restoration than stainless steel crown.
  Arms: group (1): the adaptive xp endo shaper
Procedure: pulpectomy treatment will be done using FANTA AF baby files. — the patient will be anesthetized by local anesthesia. the rubber dam will be used for isolation. caries will be removed using high speed handpiece. determination of working length using apex locator. The canal patency will be checked with a #10 K-file, and a glide path until #15 K-file will be created .the root canals of primary molars will be cleaned and shaped in pulpectomy treatment using FANTA AF baby files. it is pediatric rotary system consists of 4 files specialized for primary molars.Open file: #17, taper 08.
  * BTF1: #20, taper 04, Yellow
  * BTF2: #25, taper 04, Red
  * BTF3: #30, taper 04, Blue The file will be activated at speed 350 rpm and torque 2 N until reaching the full working length. the canals will be irrigated using 2.5% Nacol ending with 0.9% normal saline canal irrigation. the canals will be dried with paper points and obturated with Metapex. teeth will be restored by glass ionomer restoration than stainless steel crown.
  Arms: group (2): Fanta AF baby file
Procedure: pulpectomy treatment will be done using hand k files. — the patient will be anesthetized by local anesthesia. the rubber dam will be used for isolation. caries will be removed using high speed handpiece. determination of working length using apex locator. the root canals of primary molars will be cleaned and shaped in pulpectomy treatment using hand k files starting with #15 stainless steel hand K file. they are manual files, they are standard for root canal treatment (control group). the canals will be irrigated using 2.5% Nacol ending with 0.9% normal saline canal irrigation. the canals will be dried with paper points and obturated with Metapex. teeth will be restored by glass ionomer restoration than stainless steel crown.
  Arms: group (3): hand k files

SUMMARY:
The goal of this clinical trial is to compare the post operative pain after using three different instrumentation techniques in pulpectomy treatment of pediatric participant. The main question it aims to answer:

If different instrumentation techniques will affect the post operative pain in pulpectomy treatment of primary molars ? Participants will evaluate the pain using Modified Wong baker pain rating scale.

Researchers will compare [ the adaptive XP endo shaper, Fanta AF baby files, and hand K files] to see if they will affect the post operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children free from systemic diseases.
* Teeth with sufficient coronal tooth structure.
* Teeth with necrotic pulp.
* Teeth should have 2/3 of the remaining roots.

Exclusion Criteria:

* Children taking medications up to six hours before the treatment.
* Children with multiple teeth that required pulpectomy will not be included to eliminate the possibility of pain referral.
* Excessive tooth mobility.
* Teeth with perforated pulpal floor.
* Teeth with external or internal root resorption.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-05-04 (Estimated); Study Completion 2024-05-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of post-operative pain after pulpectomy treatment in primary teeth | one week
  Assessment of post-operative pain using Modified Wong-baker pain rating scale. It is 4-point scale measures pain as:
  * Score zero - no pain.
  * Score one - slight pain.
  * Score two - moderate pain. Score three - severe pain. so ( score 0 is the best score & score 3 is the worst) These data will be recorded at intervals of 6, 12, 24, 72 hours, and one week. A telephonic communication will be done with the parents by the second assessor who will be blinded to the treatment protocol at 6, 12, 72 hours to assess the pain, and the patients will be given two appointments, first after 24 hours and the second after one week from the operating day. During both visits, the second assessor will collect the results of the pain assessment from the child's parent and will cross-check all the results to ensure that the reported values are consistent.

CONTACTS AND LOCATIONS:
Locations (1):
- Amal Taha Taha Elakkad, Al Mansurah, Egypt